CLINICAL TRIAL: NCT04946123
Title: Association of Methimazole With L-carnitine and Selenium in Patients With Hyperthyroidism
Brief Title: Hyperthyroidism: Methimazole Plus L-carnitine and Selenium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-carnitine Hyperthyroidism
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methimazole (control) (No Intervention): Patients with hyperthyroidism under methimazole treatment
- methimazole+L-carnitine+selenium (intervention) (Experimental): Patients with hyperthyroidism under methimazole treatment + supplementation with L-carnitine and Selenium
  Interventions: Dietary Supplement: L-carnitine+Selenium

INTERVENTIONS:
Dietary Supplement: L-carnitine+Selenium — Supplementation with L-carnitine and Selenium
  Arms: methimazole+L-carnitine+selenium (intervention)

SUMMARY:
The study aims to investigate the benefits of methimazole treatment in patients with hyperthyroidism, associated with supplementation of L-carnitine and Selenium.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hyperthyroidism requiring therapy with methimazole

Exclusion Criteria:

* Drug and alcohol abuse;
* Pregnancy;
* Medically uncontrolled psychiatric conditions;
* Interfering therapies (lithium, interferone, TKI, amiodarone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Hyperthyroidism symptoms | Change from baseline QoL at 6 months of supplementation
  Improvement of the patients' quality of life through questionnaire
Hyperthyroidism symptoms | Change from 6-months supplementation QoL at 12 months of intervention (end of study)
  Improvement of the patients' quality of life through questionnaire

SECONDARY OUTCOMES:
TRAb | Four time points: baseline; after 3 months of supplementation; after 6 months of supplementation; end of the study (12 months)
  Change in serum TRAb (TSH receptor antibodies)
TSH | Four time points: baseline; after 3 months of supplementation; after 6 months of supplementation; end of the study (12 months)
  Change in serum TSH (Thyroid stimulating hormone)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Città della scienza e degli studi di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No